CLINICAL TRIAL: NCT00004494
Title: Phase I Study of Vasoactive Intestinal Peptide in Patients With Acute Respiratory Distress Syndrome and Sepsis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stony Brook University (Other)
Collaborators: State University of New York (Other); FDA Office of Orphan Products Development (U.S. Federal Agency)
Purpose: Treatment
Other Study IDs: 199/14275; SUNY-SB-FDR001488; SUNY-SB-96-077; SUNY-SB-98-2606; FD-R-0001488 (Other Grant/Funding Number: FDA Orphan Drug Products)
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Sepsis; Respiratory Distress Syndrome; Respiratory Distress Syndrome, Adult
Keywords: cardiovascular and respiratory diseases; immunologic disorders and infectious disorders; neonatal disorders; rare disease; respiratory distress syndrome; sepsis
MeSH Terms: conditions — Sepsis; Respiratory Distress Syndrome; Respiratory Tract Diseases; Immune System Diseases; Communicable Diseases; Infant, Newborn, Diseases; Rare Diseases | interventions — Vasoactive Intestinal Peptide

INTERVENTIONS:
Drug: vasoactive intestinal peptide

SUMMARY:
OBJECTIVES:

I. Determine the maximum tolerated dose of vasoactive intestinal peptide in patients with acute respiratory distress syndrome.

II. Evaluate the safety and pharmacodynamic activity of this peptide in these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

This is a dose escalation study.

Patients receive vasoactive intestinal peptide (VIP) IV over either 6 or 12 hours.

Cohorts of 3 patients each receive escalating doses of VIP over either 6 or 12 hours until the maximum tolerated dose is determined.

Patients are followed for 30 days.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Diagnosis of adult respiratory distress syndrome (ARDS) with sepsis

ARDS characterized by: hypoxemia refractory to supplemental oxygen therapy, diffuse pulmonary infiltrates, no cardiogenic cause of pulmonary edema, and reduced pulmonary compliance

Sepsis characterized by: Two or more of the following: Fever or hypothermia; Tachycardia; Tachypnea; WBC greater than 12,000/mm3 or less than 4,000/mm3 or immature neutrophils; Hypotension; Clinical suspicion of infection; Inadequate organ perfusion or organ dysfunction as demonstrated by: Acute deterioration in mental acuity (excluding sedatives or other nonsepsis causes) OR Unexplained metabolic acidosis OR Oliguria for greater than 2 hours OR Unexplained coagulopathy (elevated PT or PTT or platelet count decreased to less than 50% of baseline within 24 hours or less than 100,000/mm3) OR Acute elevation of bilirubin to greater than 2.0 mg/dL AND elevation of alkaline phosphatase, SGOT, or SGPT

No sepsis with unstable BP

--Prior/Concurrent Therapy--

At least 30 days since prior enrollment in investigational trial; No other concurrent enrollment in investigational trial

--Patient Characteristics--

Hematopoietic: See Disease Characteristics; No uncontrolled hemorrhage (transfusion of 4 or more units required within past 24 hours); No chemotherapy induced neutropenia (granulocyte count less than 1000/mm3)

Hepatic: No severe liver disease with portal hypertension

Renal: No anuria (urine output less than 50 mL/day)

Cardiovascular: No cardiogenic shock

Neurologic: No recent stroke, head trauma, or increased intracranial pressure; No other serious neurologic disorder

Other: Not pregnant; No acquired immune deficiency syndrome; No immunosuppressed transplant patients; No severe burns; No irreversible underlying condition with rapidly fatal course; No marked obesity; No recent history of diarrhea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 1998-09

CONTACTS AND LOCATIONS:
Overall Officials: Sami I. Said, Study Chair — State University of New York
Locations (2):
- United States (2):
  - Veterans Affairs Medical Center - Northport, Northport, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York